CLINICAL TRIAL: NCT02893514
Title: Leveraging Technology to Address Unhealthy Drug Use in Primary Care: Effectiveness of the Substance Use Screening and Intervention Tool (SUSIT)
Brief Title: Leveraging Technology to Address Unhealthy Drug Use in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-01074; 1R34DA040830-01 (NIH)
Record Dates: First submitted 2016-08-11; First posted 2016-09-08 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Addiction
Keywords: Drug Use
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening Only (SO) (Placebo Comparator)
  Interventions: Other: Screening Only (SO) condition
- Substance Use Screening and Intervention Tool (SUSIT) (Experimental)
  Interventions: Other: SUSIT Condition

INTERVENTIONS:
Other: Screening Only (SO) condition — Patient and PCP are not presented with screening results. The PCP does not receive clinical decision support, or clinical reminders.
  Arms: Screening Only (SO)
Other: SUSIT Condition — Following completion of substance use screening, the tablet computer presents screening results (including level of risk) to the patient for each substance used, asks them to identify their drug of most concern (DOMC), and assesses readiness and confidence to change behavior. Results are delivered to the PCP at the point of care, paired with clinical decision support tailored to the patient's screening results. This information is delivered on the tablet computer, which is handed to the PCP by a Medical Assistant. CDS guides the PCP through a brief intervention specific to the DOMC, recommends clinical actions pertaining to the substance and risk level, and generates a printed summary for the patient. At each scheduled follow-up medical visit, the PCP receives a clinical reminder containing a summary of the patient's substance use and level of risk, paired with CDS that guides them through a follow-up brief intervention.
  Arms: Substance Use Screening and Intervention Tool (SUSIT)

SUMMARY:
This study will develop a clinical decision support tool that assists primary care providers in carrying out substance use interventions, and then compare (in Phase 2) two clinical scenarios, screening only (SO) vs. SUSIT, (on dose of substance use brief intervention received) and changes in drug use at 3 and 6 months, among primary care patients. Investigators will develop the Clinical Decision Support (CDS) component and then test the full SUSIT approach, using mixed methods to assess its acceptability and adoption, and gathering preliminary data on its efficacy for reducing unhealthy drug use. CDS development is concurrent with the SO phase to avoid losing valuable time, but will be conducted at a secondary study site to avoid contaminating the SO condition.

DETAILED DESCRIPTION:
This study has 3 specific aims:

Aim 1 is to develop clinical decision support that assists primary care providers in carrying out a brief intervention.

Aim 2 is to assess the impact of the SUSIT on dose of substance use brief intervention received by patients.

Aim 3 is to gather preliminary evidence on the efficacy of the SUSIT approach for reducing moderate-risk drug use.

ELIGIBILITY:
Inclusion Criteria:

* Substance use screening results (collected using the tablet-based screening tool) indicating current moderate risk drug use, based on a substance specific involvement score (SSIS) indicating current (past 3 months) use of at least one drug with a moderate risk level (SSIS 4-26), in the absence of any high-risk drug or alcohol use (SSIS 27+);
* Presenting for visit with a participating PCP

Exclusion Criteria:

* Prior participation in the study (i.e. participation in the SO study phase would preclude participation in the SUSIT phase);
* Attending a formal addiction treatment program (not including informal treatment such as Alcoholics Anonymous, Narcotics Anonymous), in the past 3 months;
* Pregnant (based on self-report).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNeely, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Screening Only (SO) | Substance Use Screening and Intervention Tool (SUSIT)
Started | 42 | 37
Completed | 42 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening Only (SO) | Substance Use Screening and Intervention Tool (SUSIT) | Total
Number analyzed (Participants) | 42 | 37 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.8) | 45.0 (13.1) | 45.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 19
  Male | 27 | 33 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 10 | 9 | 19
  More than one race | 15 | 13 | 28
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 42 | 37 | 79
Clinic Type [Count of Participants; unit: Participants]
  Primary Care | 20 | 11 | 31
  HIV | 22 | 26 | 48

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Brief Intervention (BI) for Drug Use at Baseline Visit
Description: Reported by Patients
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Screening Only (SO) | Substance Use Screening and Intervention Tool (SUSIT)
Number analyzed (Participants) | 42 | 37
Participants | 17 | 33

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Screening Only (SO) | Substance Use Screening and Intervention Tool (SUSIT)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/37
Other Adverse Events (participants affected / at risk) | 0/42 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02893514/Prot_SAP_000.pdf